CLINICAL TRIAL: NCT03939858
Title: Blood-based Bioenergetic Profiling and Cognition in Glioblastoma Patients
Brief Title: Bioenergetic Profiling and Cognition in GBM Patients
Status: Terminated | Type: Observational
Why Stopped: Funding and laboratory access issues, study is closed
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00058347; NCI-2019-02984 (Other: Clinical Trial Reporting Program); WFBCCC 01219 (Other: Wake Forest Baptist Comprehensive Cancer Center)
Record Dates: First submitted 2019-05-01; First posted 2019-05-07 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Mental Status and Dementia Tests; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cognitive Function Analysis: Cognitive function will be evaluated using a customized cognitive battery designed for brain tumor patients. Tests have been selected to represent a range of cognitive functions affected by cancer and radiotherapy including basic attention, recent memory, executive functions (spanning verbal fluency, cognitive set-shifting, and abstract reasoning), and visual perceptual/spatial skills.
  Interventions: Procedure: Cognitive Assessment; Diagnostic Test: Blood Collection; Diagnostic Test: Bioenergetic Profiling

INTERVENTIONS:
Procedure: Cognitive Assessment — Tests have been selected to represent a range of cognitive functions affected by cancer and radiotherapy including basic attention, recent memory, executive functions (spanning verbal fluency, cognitive set-shifting, and abstract reasoning), and visual perceptual/spatial skills.
Diagnostic Test: Blood Collection — 16 ml of blood will be collected before 10 a.m. and after the participant has fasted for 8 hours. White blood cells and platelets will be used for respirometric analysis. Plasma will be additionally processed and saved in 500uL aliquots(x2) and the remainder in 1mL aliquots at -80°C.
Diagnostic Test: Bioenergetic Profiling — Peripheral blood mononuclear cells (PBMCs) and platelets will be separated from the blood. Primary respirometric parameters will be measured with high-throughput respirometry using the Agilent Seahorse 24XFe. Additional parameters will be collected with high-resolution respirometry using the OROBOROS Oxygraph-2k. Both methods will report a variety of mitochondrial parameters resulting in 48 measures per participant, creating robust profiles of bioenergetic health. Additional analysis will include western blots to enumerate protein density for the five major mitochondrial complexes, mtDNA copy number analysis, and citrate synthase activity as these assays provide different but complementary data to respirometry for a more dynamic picture of mitochondrial metabolism.

SUMMARY:
This trial studies the use of blood-based bioenergetic profiling and cognitive testing in assessing patients with glioblastoma undergoing chemoradiation therapy. The purpose of this pilot research study is to find out if it is possible to see changes in participants' mitochondria, parts of a cell that produce energy, that might be associated with changes in participants' brain function after chemoradiation therapy.

DETAILED DESCRIPTION:
Primary Objective:

• To determine the feasibility of performing bioenergetic profiling in glioblastoma patients receiving chemoradiation by ascertaining the proportion of patients who have enough white blood cells in a 16 mL blood to successfully perform the profiling assays.

Secondary Objectives:

• To determine if either pre-radiotherapy bioenergetic profile or the change in bioenergetic profile from pre-radiotherapy to post-radiotherapy are predictive of subacute cognitive decline after radiation.

OUTLINE: Patients undergo neurocognitive testing over 1 hour using a customized battery of tests designed for brain tumor patients at Wake Forest Baptist Comprehensive Cancer Center. Patients also undergo blood collection at baseline and at 1 and 3 months post radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

• Glioma patients greater than 18 years old receiving chemoradiation with a Karnofsky Performance Status greater than or equal to 50.

Exclusion Criteria:

* Prior diagnosis (by a physician or neuropsychologist) of any type of dementia (AD, frontotemporal dementia, vascular dementia, Lewy-body dementia, Parkinson's dementia), normal pressure hydrocephalus, Creutzfeldt Jacob disease, posterior cortical atrophy, Huntington's disease, or Korsakoff syndrome will be excluded. Patients who were diagnosed with Mild Cognitive (MCI) Impairment greater than or equal to 1 year prior to diagnosis with their high grade glioma will also be excluded. Patients reported by family members as having memory problems or with subjective memory complaints are still eligible.
* Patients taking medications known to have a mitotoxic effect (see attached appendix). Patients who take any of the as needed medications on the list more than 4 times per week will be excluded. There are medications that are considered mitotoxic that are not included on this list because of the essential nature of the medications to this population (steroids, anti-seizure medications, diabetic medications etc.) or high frequency of use in this population (statins, beta blockers).
* Patients on medications with the potential to enhance cognition including donepezil, memantine, armodafinil or methylphenidate.
* Patients who are not fluent in English will be excluded.
* Patients with aphasia or other neurologic deficit which would prevent participating in cognitive testing will be excluded.
* Patients who are unable to fast for 8 hours will be excluded since enrolled patients will only be able to drink water for the 8 hours before blood draws.
* Patients who drink more than 14 alcoholic drinks per week.
* Patients who are active smokers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Glioma patients receiving chemoradiation
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2019-10-24 (Actual); Primary Completion 2021-09-22 (Actual); Study Completion 2023-06-09 (Actual)

PRIMARY OUTCOMES:
Number of Patients Completing Bioenergetics Profiling | 3 months
  The primary outcome will be the proportion of patients who are able to have bioenergetic profiling completed at all three time points (baseline, one month after radiotherapy, three months after radiotherapy). The proportion and its 95% confidence interval will be calculated.

SECONDARY OUTCOMES:
Proportion of Participants with Decline in Cognitive Function | Three months after completion of radiotherapy
  Cognitive decline as defined as a decline from pre-radiotherapy baseline by one standard deviation on any cognitive test of memory, executive function, or attention at any time point subsequent to baseline. Cognitive function will be evaluated using a customized cognitive battery of tests designed for brain tumor patients at Wake Forest University Comprehensive Cancer Center. Each participant's raw score performance on each assessment measure will be transformed to a z-score, based on available normative data. A composite mean can then be calculated for overall performance to allow for comparison between time points. The proportion of cognitive decline at one-month and 3-month visits will be calculated.
Bioenergetics Profiling Testing - Seahorse XFe24 Analyzer | Three months after completion of radiotherapy
  High-throughput respirometry parameters will be collected to compare cognitive decline v. non-decline in participant bioenergetics profile from baseline and at each follow-up visit. The respirometry parameters will be obtained simultaneously (basal respiration, leak respiration, ATP-linked respiration, maximal respiration, spare respiratory capacity and non-mitochondrial respiration). Wilcoxon rank sum test will be used to compare pre-RT bioenergetics profile and the change in bioenergetics profile in the cognitive decline groups (decline vs. non-decline) at each follow-up visit. Simple Spearman's rank correlation coefficients will be used to relate pre-RT bioenergetics profile or change in cognitive testing to change in bioenergetics profile at each follow-up visit.
Bioenergetics Profile Testing - Oroboros O2K | Three months after completion of radiotherapy
  High-resolution respirometry parameters will be collected simultaneously to compare cognitive decline v. non-decline in participant bioenergetics profile from baseline and at each follow-up visit - (routine respiration, outer mitochondrial membrane integrity measure, fatty acid β-oxidation mediated respiration, fatty acid β-oxidation and complex I, II and glycerol-3-phosphate dehydrogenase mediated respiration, maximal electron transport chain respiration, spare respiratory capacity, maximal electron transport chain after complex I inhibition, non-mitochondrial respiration, complex IV respiration, leak respiration, complex I and II mediated maximal electron transport chain respiration and cell viability). Wilcoxon rank sum test and Simple Spearman's will be used to compare pre-RT bioenergetics profile and the change in bioenergetics profile in the cognitive decline groups (decline vs. non-decline) at each follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Cramer, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No